CLINICAL TRIAL: NCT06916923
Title: Relationship Between Dysfunctional Breathing, Exercise Capacity, and Balance in Patients With Hypertension: A Prospective Cross-Sectional Study
Brief Title: Dysfunctional Breathing, Exercise Capacity, and Balance in Hypertension
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Elif Kabasakal, LECTURER, Istinye University
Other Study IDs: ISU-2025-002
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-04

CONDITIONS: Dysfunctional Breathing; Arterial Hypertension; Exercise Capacity; Balance
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertensive Patients With Dysfunctional Breathing: Participants diagnosed with arterial hypertension who exhibit symptoms of dysfunctional breathing, as determined by the Nijmegen Questionnaire. Assessments will include anthropometric measurements, functional exercise capacity tests, and balance evaluations.

SUMMARY:
This prospective cross-sectional study aims to investigate the relationship between dysfunctional breathing (DB), exercise capacity, and balance in patients with arterial hypertension (HT). DB is characterized by abnormal breathing patterns and is associated with symptoms such as dyspnea and inefficient ventilation, regardless of the presence of organic respiratory disease. Hypertension may further exacerbate these symptoms and contribute to impaired exercise performance and postural balance. The study will assess DB using the Nijmegen Questionnaire, along with anthropometric measurements, balance tests, and functional exercise capacity evaluations. Findings may contribute to better understanding of respiratory dysfunctions in hypertensive individuals and their impact on physical performance.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years
* Diagnosed with hypertension and under follow-up for at least 6 months
* Willing to participate in the study voluntarily
* Nijmegen Questionnaire score of 23 or above

Exclusion Criteria:

* Medication change within the last month prior to study enrollment
* Presence of unstable metabolic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults aged 18 to 70 years who have been clinically diagnosed with arterial hypertension and have been under follow-up for at least six months. All participants must have a Nijmegen Questionnaire score of 23 or higher, indicating a probable presence of dysfunctional breathing. Individuals must be willing to voluntarily participate in the study. Participants with recent medication changes (within the past month) or with unstable metabolic diseases will be excluded.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Assessment of Dysfunctional Breathing Level | At baseline
  Nijmegen Questionnaire: The questionnaire is used for the assessment and identification of respiratory dysfunction, unexplained respiratory symptoms, and hyperventilation syndrome indicators. It consists of 16 items covering neurological, cardiovascular, respiratory, gastrointestinal, and psychological factors. Each item is rated on a 5-point Likert scale, with a total score ranging from 0 to 64. Higher scores indicate an increased likelihood of respiratory dysfunction and hyperventilation syndrome. A score above 23 supports the possible diagnosis of dysfunctional breathing. The questionnaire has a sensitivity of 91% and a specificity of 95%. The Turkish version of the questionnaire has been validated and found to be reliable.
Assessment of Balance-I | At baseline
  The Timed Up and Go Test is a method used to rapidly assess an individual's balance control. During the test, the participant is instructed to rise from a seated position in a chair, walk a distance of 3 meters, turn around a reference object, return to the chair, and sit down again. The time taken to complete the task is recorded in seconds. The test will be repeated three times, and the average of the three trials will be used for analysis.
Assessment of Balance-II | At baseline
  The Berg Balance Scale is used to assess balance through progressively challenging tasks by reducing the level of support provided by the surface. The scale consists of 14 items, each scored from 0 to 4 (4: best performance, 0: poorest performance). A total score between 41-56 indicates a low risk of falling, 21-40 reflects a medium fall risk, and scores below 20 indicate a high fall risk.
Neck Circumference Measurements | At baseline
  Neck circumference will be measured using a flexible plastic measuring tape at the level of the cricoid cartilage, with the participant in an upright and relaxed position
Waist Circumference Measurement | At baseline
  Waist circumference will be measured using a flexible plastic measuring tape at the level of the iliac crest, with the participant standing upright and breathing normally.

CONTACTS AND LOCATIONS:
Overall Officials: Kabasakal, Study Chair — Istinye University
Locations (1):
- Istınye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP